CLINICAL TRIAL: NCT06332898
Title: The Effects of a Nutritional Supplement on Nutrient Status and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Athletic Greens International (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AG-01-0324
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Nutrition, Healthy; Gastrointestinal Microbiome; Healthy Aging

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo Controlled Design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Maltodextrin + Flavoring
  Interventions: Dietary Supplement: Placebo
- AG1 - Nutritional Supplement (Experimental): AG1, a foundational nutritional supplement
  Interventions: Dietary Supplement: AG1 - Nutritional Supplement

INTERVENTIONS:
Dietary Supplement: AG1 - Nutritional Supplement — A foundational nutritional supplement consisting of vitamins, minerals, probiotics, prebiotics, and whole food ingredients
  Arms: AG1 - Nutritional Supplement
Dietary Supplement: Placebo — Maltodextrin placebo
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled study of N=120 apparently healthy men and women. The purpose of this study is to assess the effect of a novel dietary supplement on blood markers of nutrient status, gut microbiome, and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Provide voluntary signed and dated informed consent.
* No known history of chronic illness or disease.
* Aged between 18 and 59.9 years (inclusive).
* Body Mass Index of 20-34.9 (inclusive).
* Willing to duplicate their previous 24-hour diet, refrain from caffeine and exercise for 24 hours, and fast for 10 hours prior to each Quest visit.
* Agree to maintain existing dietary and physical activity patterns throughout the study period.
* Willing and able to comply with the study protocol.

Exclusion Criteria:

* History of unstable or new-onset cardiovascular, liver, or renal conditions.
* History of diabetes or endocrine disorder.
* Multivitamin/Multimineral supplement consumption within the past 3 months.
* Regular consumption (i.e., at least five days/week) of resveratrol, quercetin, pterostilbene, coQ10, grapefruit, nicotinamide riboside, probiotics, prebiotic fiber, green tea, niacin (vitamin B3), or products meant to promote "healthy aging" or "anti-aging" or "longevity" in the 2 months prior to screening as well as throughout the study.
* Subjects who have received an antibiotic, antifungal, antiparasitic, or antiviral treatment within 90 days prior to study.
* History of use of medications or dietary supplements known to confound the study or its endpoints.
* Excessive alcohol consumption (more than 2 standard alcoholic drinks per day or more than 10 drinks per week) or drug abuse or dependence within the past 6 months.
* Current smokers or smoking within the past month.
* History of hyperparathyroidism or an untreated thyroid condition.
* History of malignancy in the previous 5 years except for non-melanoma skin cancer (basal cell cancer or squamous cell cancer of the skin).
* Prior gastrointestinal bypass surgery (Lapband, etc.).
* Other known gastrointestinal or metabolic conditions that might impact nutrient absorption or metabolism, e.g., short bowel syndrome, IBS/IBD, diarrheal illnesses, history of colon resection, gastroparesis, Inborn errors of metabolism (such as PKU).
* Chronic inflammatory condition (e.g., rheumatoid arthritis, Crohn's, ulcerative colitis, Lupus, HIV/AIDS, etc.).
* Previous medical diagnosis of asthma, gout, or fibromyalgia.
* Pregnant women, women trying to conceive, women less than 120 days postpartum, or nursing women.
* A change in hormone therapy, including oral contraceptives, within 4 weeks prior to screening, or unwilling to maintain current hormone therapy/oral contraceptive use throughout the course of the study.
* Known allergy or sensitivity to any ingredient in the test formulations as listed in the product label.
* Currently participating in another research study with an investigational product or have been in another research study in the past 30 days.

>10% weight change in the last 6 months.

- Specific exclusion type diets like vegan, vegetarian, carnivore, paleo, atkins, ketogenic etc.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2024-03-31 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Homocysteine | 90 days
  Circulating Serum Homocysteine Concentrations (umol/L)
Vitamin B12 | 90 days
  Circulating Serum Vitamin B12 Concentrations (pg/mL)
Folate | 90 days
  Circulating Serum Folate Concentrations (ng/mL)
Red Blood Cell Folate | 90 days
  Circulating Red Blood Cell Folate Concentrations (nmol/L)
Zinc | 90 days
  Circulating Serum Zinc Concentrations (ug/dL)
Vitamin C | 90 days
  Serum Vitamin C Concentrations (
Gut Microbiome | 90 days
  Examine changes in the gut microbiome structure and function measured by shallow shotgun metagenomics. Examine enrichment of taxa and metabolic pathways in the gut microbiome as a result of dietary supplementation.

SECONDARY OUTCOMES:
Dietary habits | 90 Days
  Automated Self-Administered 24-Hour (ASA24®) Dietary Assessment Tool
Gastrointestinal Health | 90 Days
  Gastrointestinal symptom rating scale (GSRS). Symptom score change after 90 days of administration, compared to Baseline. Score base on a 1-7 scale with a higher score meaning a worse outcome.
Fatigue & energy | 90 Days
  Multidimensional Fatigue Inventory (MFI).The MFI is a 20-item instrument consisting of several subscales including general fatigue and reduced activity and will be assessed after 90 days of administration compared to baseline.
Well-being | 90 Days
  World Health Organization-5 Well-being Index Questionnaire.The World Health Organization-5 Well-Being Index is a brief scale, composed of five questions in which the participants indicate in each one of them, based on the last two weeks, the frequency of their sensations, being 0 (at no time) and 5 (all of the time). The result is given as the sum of the numbers of each statement, with values ranging from 0, which represents the worst possible quality of life and 25, which is associated with the best possible quality of life. Will be assessed at baseline and after 90 days of administration.
Complete Metabolic Blood Panel | 90 Days
  Serum concentrations of sodium, potassium, carbon dioxide, chloride, albumin, total protein, glucose, and calcium., ALT, AST, bilirubin, BUN, creatinine
Complete Blood Count | 90 Days
  Circulating concentrations of white blood cells, red blood cells, hemoglobin, and hematocrit

CONTACTS AND LOCATIONS:
Overall Officials: Ellen O'Gorman, Principal Investigator — Citruslabs
Locations (1):
- Citruslabs, Santa Monica, California, United States